CLINICAL TRIAL: NCT05698134
Title: Rotational Thromboelastometry (ROTEM™) Guided Transfusion for Elective Procedures in Patients With Cirrhosis (REduCe): An Open Label Randomized Controlled Trial.
Acronym: REduCe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/3087
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cirrhosis, Liver
Keywords: ROTEM; Invasive Procedure; Cirrhosis; Blood Product
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups:
  First group will receive standard of care based on institutional protocol for blood product transfusion Second group will receive ROTEM guided protocol for blood product transfusion
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Participants will receive blood products transfusion based on prevailing institution protocol, which is based on Platelet count and coagulation parameters (APTT, PT/INR)
  Interventions: Other: Standard of care
- ROTEM guided Group (Experimental): Participants will receive blood products transfusion based on ROTEM results
  Interventions: Diagnostic Test: ROTEM

INTERVENTIONS:
Diagnostic Test: ROTEM — ROTEM is a commercially available whole blood Viscoelastic-Haemostatic Assay(VHA) point-of-care, global and dynamic haemostasis assessment tests that measures the viscoelastic changes occurring during the haemostatic process. They provide real-time, comprehensive reflection of the interaction between plasma, blood cells and platelets. It display hypo or hyper-coagulable features in patients with cirrhosis. It is widely used prior to cardiac, obstetric, trauma and liver transplant surgery to assess and correct for coagulation defects.
  Arms: ROTEM guided Group
Other: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
REDuCe is designed to evaluate the role of ROTEM™ in determining the need and the amount of pre-emptive blood products use in patients with cirrhosis undergoing elective procedures compared to the current standard of care. The secondary aim of this study is to evaluate ROTEM™ parameters in patients with acute decompensation, acute on chronic liver failure and acute liver failure and to co-relate it with the conventional coagulation tests.

DETAILED DESCRIPTION:
Patients with cirrhosis who meets eligibility criteria will be divided into two groups

1. Those who are undergoing elective procedures will be randomized into 1:1 ratio into either standard of care (institutional transfusion protocol) or ROTEM guided protocol. Baseline ROTEM will be obtained before and after blood product transfusion.
2. Those who are not for elective procedures and does not meet criteria for randomization will be entered into data collection for secondary endpoints analysis. These patients will have baseline ROTEM before transfusion and post transfusion ROTEM in those who require blood prodducts transfusion.

ELIGIBILITY:
Inclusion Criteria:

Patients with Cirrhosis undergoing elective procedure must meet all following criterias.

1. Patients undergoing the following elective procedures will be included in the study

   1. Gastroscopy with endoscopic variceal ligation
   2. Colonoscopy with polypectomy and endoscopic mucosal resection
   3. ERCP with sphincterotomy
   4. Percutaneous liver biopsy
   5. Biopsy of other sites (excluding liver)
   6. Hepatic venous pressure gradient with or without liver biopsy
   7. Elective Transjugular Intrahepatic Portosystemic Shunt
   8. Portal Vein embolization
   9. Trans-arterial chemo-embolization (TACE)
   10. Thermal ablation of hepatocellular carcinoma
   11. Large volume paracentesis
   12. Central venous catheter insertion
   13. Thoracentesis
2. Age: Older than 21 years
3. Coagulopathy based on conventional coagulation tests which is defined as

   1. INR > 1.5 and/or aPTT > 1.5x ULN for PTT and/or
   2. Platelets < 50,000/mm3/uL
4. Patients with acute decompensation, acute on chronic liver failure and acute liver failure.
5. Able to give informed consent.

Exclusion Criteria:

1. Emergency procedures. (defined as life-saving procedures)
2. On-going bleeding
3. Under 21 years of age
4. Inability to obtain informed consent from patients
5. Coagulation disorders (other than those relating to liver disease)
6. Patients on anticoagulant medications (e.g. warfarin, enoxaparin, rivaroxaban, dabigatran, apixaban, heparin, clexane etc.)
7. Patients on anti-platelet aggregation agents other than aspirin (e.g. clopidogrel, ticagrelor)
8. Active malignancy except hepatocellular carcinoma
9. Patients who have received FFP, platelet transfusion, cryoprecipitate within last 7 days
10. Patients with stage 4 or 5 chronic kidney disease
11. Patients receiving renal replacement therapy
12. Patients with active sepsis as defined by ACPP-SCCM criteria (21).
13. Pregnant Women

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-28 (Estimated); Study Completion 2023-05-28 (Estimated)

PRIMARY OUTCOMES:
Difference in amount of blood products transfused | 24 months
  The difference in amount/volume of blood products used(fresh frozen plasma in mls, cryoprecipitate in units and platelets in units) used in patients with cirrhosis undergoing elective procedure.

SECONDARY OUTCOMES:
Peri-procedural bleeding complications | 24 months
  1. Peri-procedural bleeding complications (e.g. immediate, and delayed bleeding) defined as overt bleeding or haemoglobin drop requiring transfusion with a target of 8 g/dL.
  1. Immediate Bleeding (<24 hours of procedure)
  2. Delayed bleeding (> 24 hours of procedure)
Transfusion related adverse events | 24 months
  Adverse events are defined as any side effect occurring within 6 hours of blood product infusion
Hospital Length of stay | 24 months
  Total hospital length of stay (in days)
30-day and 90-day survival | 24 months
  Survival rate at 30-day and 90-day from time of procedure
Thrombotic Complications | 24 months
  Thrombotic events such as portal vein thrombosis, stroke which may be secondary to blood product transfusion
Procedure related complications-other than bleeding | 24 months
  Non-bleeding related complications, specific to procedure such as pneumothorax will be reviewed

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar R, Ng LXL, Wong YJ, Tan CK, Wang LZ, Qiu TY, Wong B, Lin KW, Li JW, Kwek ABE, Ang TL, Gokhle RS, Sivanath TP. Rotational Thromboelastometry Reduces the Need for Preemptive Transfusion in Cirrhosis: A Randomized Controlled Trial (NCT:05698134). J Clin Exp Hepatol. 2025 Jan-Feb;15(1):102409. doi: 10.1016/j.jceh.2024.102409. Epub 2024 Sep 7. PMID 39391324